CLINICAL TRIAL: NCT02122757
Title: Randomised Sham-controlled Trial of Anodal Transcranial Direct Current Stimulation (tDCS) for the Prevention of Episodic Migraine
Brief Title: Anodal Transcranial Direct Current Stimulation of the Visual Cortex Versus Sham Stimulation in the Episodic Migraine
Acronym: ANODEM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean Schoenen, Honorary Full Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CB-1300
Record Dates: First submitted 2013-11-04; First posted 2014-04-25 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Sporadic Migraine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Anodal Cefaly tDCS (Placebo Comparator): 2 mA placebo anodal tDCS (the direct current is delivered just for 30 seconds) is applied over the visual cortex for 20 minutes, everyday for 2 months, in 15 patients
  Interventions: Device: sham Cefaly tDCS
- Anodal Cefaly tDCS (Active Comparator): 2 mA anodal tDCS is delivered over the visual cortex, for 20 minutes, everyday for 2 months, in 15 patients.
  Interventions: Device: Cefaly tDCS

INTERVENTIONS:
Device: Cefaly tDCS — Cefaly tDCS (transcranial direct current stimulation) is able to modify cortical excitability, in particular anodal tDCS increases it. The side effects of tDCS are minor, especially sensations of itching and scalp paresthesias.
  Arms: Anodal Cefaly tDCS
Device: sham Cefaly tDCS — 2mA during 30sec
  Arms: Sham Anodal Cefaly tDCS

SUMMARY:
Anodal tDCS increases the excitability of the cerebral cortex and its daily application during intercritical phase, may have a therapeutic effect in episodic migraine.

DETAILED DESCRIPTION:
During the interictal phase, the cerebral cortex is characterised by hyperresponsiveness to repeated sensory stimuli, manifested by a lack of habituation or adaptation of cortical evoked responses. Such habituation deficit can be shown in the visual cortex by the study of visual evoked potentials (VEP) and it is possibly explained by a reduction in the cortical pre-activation level due to thalamo-cortical dysrhythmia. In healthy subjects and in migraineurs between attacks, anodal tDCS increases VEP habituation and 1st block amplitude. In a proof-of-concept trial, the investigators have shown in 10 episodic migraine without aura patients that 2 weekly 15-minute sessions for 8 weeks of anodal tDCS over the visual cortex significantly decreased attack frequency, migraine days, attack duration and acute medication intake for more than 4 weeks after the last treatment session.

This randomized trial was designed to prove the preventive effect in episodic migraine of anodal tDCS over the visual cortex compared to sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of episodic migraine with (ICHD III beta 1.2.1) or without aura (ICHD III beta 1.1)

Exclusion Criteria:

* preventive treatment
* others diseases or contraindications to tDCS (epilepsy, pacemaker, metal prosthetics)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Migraine frequency | 6 months
  The investigators evaluate the migraine frequency at baseline (2 months), during the treatment and 2 months after its end.

SECONDARY OUTCOMES:
Migraine intensity | 6 months
  The investigators evaluate migraine intensity at baseline, during the treatment and 2 months after its end.
Acute medication intake | 6 months
  The investigators evaluate acute medication intake at baseline, during the treatment and 2 months after its end.
Attack duration | 6 months
  The investigators evaluate attack duration at baseline, during the treatment and 2 months after its end.
Score on psychological scales | 6 Months
  The investigators evaluate score on psychological scales at baseline, during the treatment and 2 months after its end.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Magis, MD,PhD, Principal Investigator — University of Liege; Jean Schoenen, MD,PhD, Study Director — University of Liege
Locations (1):
- Roberta Baschi, Liège, Belgium